CLINICAL TRIAL: NCT00728338
Title: Effect of Docosahexenoic Acid (22:6n-3, DHA) Supplementation on Risk Factors for Cardiovascular Disease in Hyperlipidemic Men
Brief Title: Docosahexenoic Acid (DHA) Supplementation and Cardiovascular Disease in Men With High Triglycerides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: VA Northern California Health Care System (U.S. Federal Agency); DSM Nutritional Products, Inc. (Industry)
Responsible Party: Darshan S. Kelley, Ph.D., USDA, ARS, WHNRC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WHNRC002
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Hypertriglyceridemia
Keywords: docosahexenoic acid (DHA); dietary supplement; n-3 polyunsaturated fatty acid; cardiovascular disease
MeSH Terms: conditions — Hypertriglyceridemia; Cardiovascular Diseases | interventions — Docosahexaenoic Acids; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Martek Biosciences Corporation Neuromins Capsules 7.5 g DHA oil/day
  Interventions: Dietary Supplement: Docosahexenoic acid (DHA)
- 2 (Placebo Comparator): 7.5 g/ day olive oil
  Interventions: Dietary Supplement: Olive oil

INTERVENTIONS:
Dietary Supplement: Docosahexenoic acid (DHA) — The DHA group received 7.5 g/d DHA oil (DHA 3.0 g/d) which is produced in the microalga Crypthecodinium cohinii.
  Other Names: Martek Biosciences Corporation, Neuromins Capsules
  Arms: 1
Dietary Supplement: Olive oil — 7.5 g olive oil/day
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effects of supplementing diets of hyperlipidemic men with DHA (docosahexenoic acid) on risk factors for cardiovascular disease. We hypothesize that supplementing diets of hyperlipidemic men with DHA will decrease the plasma concentrations of CRP (C-reactive protein), inflammatory cytokines, and soluble adhesion molecules. We further hypothesize that DHA supplementation will decrease serum triglyceride concentrations and increase HDL concentration.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) and stroke are the leading causes of mortality in the United States, accounting for more than 38% of all deaths. Elevated total- and LDL- cholesterol, number of total and small dense LDL particles, triacylglycerols, and low HDL-C are established independent risk factors for the development of CVD. Additional novel blood lipid markers used as risk factors for CVD include, increased plasma concentration of remnant like particle-cholesterol (RLP-C), decreased ratio between plasma eicosapentaenoic acid (EPA) and arachidonic acd (AA), and decreased omega-3 index (sum of EPA and DHA as a percentage of total fatty acid content) of the red blood cells.

Diets rich in omega-3 fatty acids have been shown to be cardio-protective; these diets decreased inflammation, platelet aggregation, cardiac arrhythmias, triglycerides, number of total LDL and small dense LDL particles, and increased omega-3 index, endothelial relaxation and atherosclerotic plaque stability. Most of the earlier studies regarding the effects of long chain n-3 PUFA on blood lipids were conducted with fish oils which contain a mixture of EPA and DHA. Recently a number of studies have been conducted with EPA and DHA individually. Results from studies with individual fatty acids show that EPA and DHA have similar effects on some of the lipid parameters, but they are assimilated to a different concentration in tissues and have different effects on lipoprotein particle size, heart rate and blood pressure. The main purpose of this study is to examine the effects of DHA supplementation on the above three risk factors.

ELIGIBILITY:
Inclusion Criteria:

* fasting serum triglyceride values of 150-400 mg/dL
* total cholesterol < 300 mg/dL
* LDL-cholesterol < 220 mg/dL
* BMI between 22 and 35 Kg/m2

Exclusion Criteria:

* anti-inflammatory medications including steroids
* antihypertensives
* non sulfonyl urea medications for diabetes mellitus
* drugs that alter serum triacylglycerols and HDL-C levels (i.e. fibrates)
* niacin supplements
* consumers of illegal substances
* consumers of more than 5 drinks of alcohol per week
* more than one fish meal per week
* dietary supplements of fish oil, flaxseed oil or vitamin C or E

Ages: 39 Years to 66 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-06; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Plasma biomarkers of inflammation | 0, 45, and 90 days

SECONDARY OUTCOMES:
Granulocyte maturation | 0, 45, and 90 dyas
fasting and post-prandial serum lipids and lipoproteins | 0, 45, and 90 days
blood pressure and blood clotting | 0, 45, and 90 days
plasma biomarkers for diabetes | 0, 45, and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Darshan S Kelley, PhD, Principal Investigator — USDA, ARS, WHNRC
Locations (1):
- Usda, Ars, Whnrc, Davis, California, United States

REFERENCES:
- [Result] Kelley DS, Siegel D, Vemuri M, Mackey BE. Docosahexaenoic acid supplementation improves fasting and postprandial lipid profiles in hypertriglyceridemic men. Am J Clin Nutr. 2007 Aug;86(2):324-33. doi: 10.1093/ajcn/86.2.324. PMID 17684201
- [Result] Kelley DS, Siegel D, Vemuri M, Chung GH, Mackey BE. Docosahexaenoic acid supplementation decreases remnant-like particle-cholesterol and increases the (n-3) index in hypertriglyceridemic men. J Nutr. 2008 Jan;138(1):30-5. doi: 10.1093/jn/138.1.30. PMID 18156400
- [Derived] Kelley DS, Adkins Y, Woodhouse LR, Swislocki A, Mackey BE, Siegel D. Docosahexaenoic acid supplementation improved lipocentric but not glucocentric markers of insulin sensitivity in hypertriglyceridemic men. Metab Syndr Relat Disord. 2012 Feb;10(1):32-8. doi: 10.1089/met.2011.0081. Epub 2011 Oct 14. PMID 21999398
- [Derived] Dawson K, Zhao L, Adkins Y, Vemuri M, Rodriguez RL, Gregg JP, Kelley DS, Hwang DH. Modulation of blood cell gene expression by DHA supplementation in hypertriglyceridemic men. J Nutr Biochem. 2012 Jun;23(6):616-21. doi: 10.1016/j.jnutbio.2011.03.004. Epub 2011 Jul 19. PMID 21775114
- See also: USDA, ARS, WHNRC — http://www.ars.usda.gov/main/site_main.htm?modecode=53062500